CLINICAL TRIAL: NCT07271173
Title: Study on the Effects of Unilateral Resistance Training on Lower Limb Muscle Strength and Symmetry After Anterior Cruciate Ligament Reconstruction Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M2025001
Record Dates: First submitted 2025-11-20; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-10

CONDITIONS: Anterior Cruciate Ligament Reconstruction Rehabilitation
MeSH Terms: interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group: Bilateral resistance training group (Active Comparator): Control group: Bilateral resistance training (BRT, referring to the training method where both limbs (both hands or both legs) simultaneously resist the same resistance. The force is transmitted synchronously on both sides, the center of gravity is stable, and the movements are symmetrical). The movements in the BRT group were similar to those in the URT group. Each movement was completed simultaneously by both legs. The resistance setting was based on measuring the 1RM of both lower limbs (60% of 1RM).
  Interventions: Behavioral: resistance training
- Experimental group: Unilateral resistance training group (Experimental): Experimental group: Unilateral Resistance Training (URT, referring to the training method where one limb (either one hand or one leg) performs resistance movements independently, emphasizing the application of load to the target limb while activating the stabilizing muscle groups on the opposite side to maintain balance). In the URT group, each movement is performed first by the affected leg and then by the healthy leg. A set is completed when both legs have finished. After the training of the affected leg, the timing begins. The training time of the healthy leg also counts as the interval time. The resistance setting is measured separately for each side of the lower body's single side (1RM) at 60% of 1RM.
  Interventions: Behavioral: resistance training

INTERVENTIONS:
Behavioral: resistance training — After signing the informed consent form, the relevant indicators for the pre-trial tests can be conducted.Outcome assessments are conducted at baseline (1 day before the intervention) and 3 days after the final training session (day 45 of the study).The entire trial period lasts for 6 weeks, with 3 training sessions per week. The entire training process includes 5 minutes of warm-up (power bike), 5 minutes of core strength training, 50 minutes of muscle strength training, and 10 minutes of stretching training. The training methods of the two groups are only different in the muscle strength training method. The experimental group (URT group) performs unilateral resistance training for both lower limbs, while the control group (BRT group) performs bilateral resistance training for both lower limbs. There are a total of 6 training actions: towel roll compression training, sitting leg-cranking training, knee extension resistance training, distant hip bridge train

SUMMARY:
Brief Summary Study type: Randomized controlled trial (interventional). Purpose: To find out whether six weeks of unilateral resistance training (URT) improves lower-limb strength and inter-limb symmetry more than traditional bilateral resistance training (BRT) after anterior cruciate ligament reconstruction (ACLR).

Main questions:

Does URT produce better limb-symmetry in knee flexor/extensor peak torque than BRT? Does URT lead to larger gains in feed-forward motor control, Lysholm knee score and International Knee Documentation Committee 2000 (IKDC 2000) subjective rating? Comparison: Participants will be randomly assigned to URT (each exercise done one leg at a time) or BRT (both legs work together). Training volume, frequency, session length and progression rules are identical in both groups.

What participants will do: After giving consent, complete baseline tests of strength, motor control and knee questionnaires. Attend 3 supervised sessions per week for 6 weeks. Each session lasts ~70 min:

5 min warm-up on cycle ergometer 5 min core-stability work 50 min strength circuit (6 exercises, 2 min between sets, 3 min between exercises) 10 min stretching/cool-down One-repetition maximum (1RM) re-tested at week 3 to adjust load. Final assessment within 3 days after the last training session (same tests as baseline).

DETAILED DESCRIPTION:
Detailed Description This single-center, prospective, randomized controlled trial will enroll 48 patients who have undergone primary anterior cruciate ligament reconstruction (ACLR) at Chongli Campus, Peking University Third Hospital. After providing written informed consent, participants will be randomly allocated in a 1:1 ratio to either the unilateral resistance training (URT) group or the bilateral resistance training (BRT) group (24 per group).

URT: Each exercise is performed independently with one limb at a time, isolating the target limb while contralateral stabilizers are simultaneously activated to maintain balance.

BRT: Both limbs simultaneously move against a shared resistance, keeping the center of gravity stable and the movement symmetrical.

Baseline assessments will be completed within one week before the first training session; post-intervention testing will occur within three days after the final session. The program lasts six weeks, with three supervised sessions per week. Every session comprises:

5-min warm-up on a cycle ergometer 5-min core-stability work 50-min strength training (the only component that differs between groups) 10-min stretching and cool-down Six exercises are prescribed in identical order for both groups: towel-squeeze press, seated leg press, knee-extension against resistance, long-lever glute bridge, prone hamstring curl, and Romanian dead-lift. Two minutes of rest are given between sets; three minutes separate exercises. Load is set at 60 % of the relevant one-repetition maximum (1RM), re-tested at baseline and week 3 to allow progression.

URT protocol: Each exercise is executed first by the involved leg, then immediately by the uninvolved leg; completion of both sides constitutes one set. The time needed for the uninvolved leg is counted as part of the inter-set interval.

BRT protocol: Both legs work simultaneously; 1RM is determined bilaterally. Training volume, frequency, session duration, and progression criteria are therefore identical; only the resistance modality (unilateral vs bilateral) differs.

Primary outcomes are limb-symmetry indices for peak torque of knee extensors and flexors (isokinetic dynamometry). Secondary endpoints include feed-forward motor control scores, Lysholm knee scale, and IKDC 2000 subjective evaluation. All measurements are obtained pre-intervention and at week 6. The study will determine whether six weeks of URT confers superior strength recovery and inter-limb symmetry compared with conventional BRT after ACLR.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-55 years
* ACLR performed with hamstring-tendon autograft ≥ 3 months ago
* Full extension (no loss) and ≤ 5° difference in knee-flexion range between limbs, with flexion ≥ 120°
* Able to recruit quadriceps adequately (no lag during 10 consecutive straight-leg raises on the involved side)
* Can stand pain-free on the involved leg for ≥ 5 s without support
* Has signed informed consent and can complete all study procedures

Exclusion Criteria:

* Previous lower-limb surgery on either leg, including revision ACLR
* Any prior knee surgery on the contralateral limb
* Associated ligament ruptures or fractures
* Severe patellar chondral damage
* Post-operative arthrofibrosis
* Professional athletes
* Cardiac disease
* Pregnant or lactating women

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2025-04-06 (Actual); Primary Completion 2025-11-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
muscle strength | Baseline (1 day before the intervention) and 3 days after the final training session (day 45 of the study)
  Isokinetic muscle strength test Before the test, the participants were instructed on the basic principles of isokinetic strength testing and were required to perform three maximum knee extensions as a warm-up. After the warm-up, the patients rested for 2 minutes, and then performed 5 repetitions at speeds of 60°/s and 180°/s. The peak torque values (PT) of the quadriceps and hamstring muscles of both limbs during the 5 attempts were recorded.

SECONDARY OUTCOMES:
Thigh circumference measurement (unit: cm) | Baseline (1 day before the intervention) and 3 days after the final training session (day 45 of the study)
  The patient lies on their back, in a relaxed position, with both legs naturally apart. The tape measure is placed 10 cm above the upper edge of the patella and measures the length for one week. (During the measurement, the tape measure should be firmly attached to the skin, not too tight or too loose.) Measurements are taken three times on each side, and the average value is calculated, accurate to one decimal place.
Lysholm knee score scale | Baseline (1 day before the intervention) and 3 days after the final training session (day 45 of the study)
Knee joint IKDC 2000 score | Baseline (1 day before the intervention) and 3 days after the final training session (day 45 of the study)
Single-leg jump (unit: cm) | Baseline (1 day before the intervention) and 3 days after the final training session (day 45 of the study)
  Single-leg jump (unit: cm):
  The patient places both hands behind their back and performs a single-leg jump. Measure three times and take the farthest distance. The patient is instructed to start from the uninjured leg and place their toes behind the marked starting line. Use a standard tape measure to measure the jumping distance from the starting line to the patient's heel. The measurement can be taken only if the patient can remain stable after landing; otherwise, the measurement needs to be redone.
Landing Error Scoring System,LESS | Baseline (1 day before the intervention) and 3 days after the final training session (day 45 of the study)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital of Chongli, Zhangjiakou, Hebei, China

IPD SHARING:
Plan to Share IPD: No